CLINICAL TRIAL: NCT06556550
Title: Stereotactic Radiation Therapy for Oligometastasis (1-5) in Various Tumor Sites in Comparison to Palliative Care of Oligometastatic Tumors.
Brief Title: Stereotactic Radiotherapy for Oligometastasis (1-5) in Various Tumor Sites vs. Palliative Care
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Medical Research Radiological Centre of the Ministry of Health of Russia (Other)
Responsible Party: Principal Investigator, Konstantin Gordon, Senior Researcher, National Medical Research Radiological Centre of the Ministry of Health of Russia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024_40_3
Record Dates: First submitted 2024-08-08; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Oligometastatic Disease
Keywords: stereotactic radiation therapy; stereotactic body radiation therapy; stereotactic ablative radiation therapy; Oligometastatic Disease
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic Ablative Radiotherapy (SABR) arm (Experimental): The method of stereotactic radiation therapy in patients with oligometastatic forms of tumors of various localizations after the current line of chemotherapy T1-4, N0-3, M0-1, aged over 18 years at the time of initiation of treatment
  Interventions: Radiation: stereotactic ablative radiation therapy
- Standart care arm (Active Comparator): Palliative radiation therapy or chemotherapy alone in patients with oligometastatic forms of tumors of various localizations after the current line of chemotherapy T1-4, N0-3, M0-1, aged over 18 years at the time of initiation of treatment
  Interventions: Radiation: palliative radiation therapy; Drug: Chemotherapy

INTERVENTIONS:
Radiation: stereotactic ablative radiation therapy — stereotactic ablative radiation therapy in effective doses to each metastatic site
  Arms: Stereotactic Ablative Radiotherapy (SABR) arm
Radiation: palliative radiation therapy — palliative radiation therapy (8 Gy/1 Fx, 3 Gy x 10-15 Fx, 4,5 Gy x 5 Fx)
  Arms: Standart care arm
Drug: Chemotherapy — prescribed drug line
  Arms: Standart care arm

SUMMARY:
Currently, the usual standard of palliative treatment used in patients with diagnosed oligometastatic cancer in accordance with the local clinical recommendations is chemotherapy and/or a symptomatic course of radiation therapy in doses less than ablative ones The aim of the study is to increase the effectiveness of treatment of patients with tumors of various localizations with oligometastases in the bones and internal organs with the help of stereotactic radiation therapy.

The method of stereotactic radiation therapy will be applied in patients with oligometastatic forms of tumors of various localizations after the current line of chemotherapy treatment T1-4, N0-3, M0-1, over 18 years of age at the start of treatment, compared with standard methods of palliative therapy in those same patient models.

DETAILED DESCRIPTION:
1. A patient with a previously verified diagnosis of a malignant neoplasm of one of the localizations (ICD 10-11 codes С18, С19, С20, С34, С50, С61, С64) who meets the inclusion criteria, after randomization by random numbers into the study group, is carried out:

1. 3-dimensional/4-dimensional computed tomography for simulation using specialized fixation devices (the choice of the method of computed tomography and fixing devices will be carried out depending on the location of the metastasis).
2. The resulting images are added to the contouring program.
3. Delineation of targets and risk organs is performed.
4. The clinical volumes and margins for the errors are determined.
5. Prescribing the total dose per target and dose limits for critical structures.
6. Dosimetric planning of the course of external-beam radiation therapy is carried out.
7. Irradiation sessions are carried out on a linear accelerator with a multi-leaf collimator, with the presence of a function for visual control of the target using cone tomography with a kilo-voltage/mega-voltage beam.
8. When the target is localized in the lungs, liver, and adrenal glands, in order to reduce the radiation load on the surrounding healthy tissues and achieve the necessary control over the position of metastasis, irradiation is carried out with a deep breath hold, or at certain phases of respiration.

Tumor localization / Description /Total focal dose, Gy/ Number of fractions /Single focal dose, Gy/ Irradiation mode:

Lung Tumors:

1. of 3cm or less located in the parenchyma TD45Gy in 3Fx with 15Gy every day
2. adjacent to the chest wall or less than 3 cm TD50Gy in 5Fx with 10Gy every day
3. within 2 cm of the mediastinum or brachial plexus TD60Gy in 8Fx with 7.5Gy every day

Bones TD24Gy in 3Fx with 8Gy every day

Brain Metastasis

1. volume from 0.5 to 5 cm3 TD20-22Gy in 1Fx at a time
2. volume of metastasis is from 5 to 10 cm3 TD16-18Gy or TD18-20Gy in 1 Fx at a time

Liver Radiation regimen selection based on tolerance of surrounding tissues and diligence to critical structures TD30-60Gy in 3-8Fx with 6-15Gy every day

Adrenal Glands TD60Gy in 8Fx with 7.5Gy every day

2. The expected duration of the patient's participation in clinical testing, a description of the sequence and duration of all periods of clinical testing, including the period of follow-up, if any;

Periods of clinical testing:

* pre-hospital (includes a comprehensive examination of the patient before treatment)
* inpatient (includes pre-radiation training for up to 3 working days, remote radiation therapy, from one to eight working days);
* follow-up - after 3, 6, 9, 12, 18, 24 months;
* collection and processing of the received data.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed malignant formation (ICD 10-11 codes С18, С19, С20, С34, С50, С61, С64).
2. 0-2 points on the WHO/ECOG scale of assessment of the general condition of the patient.
3. The absence of disease progression after the current line of chemotherapeutic treatment.
4. The number of oligometastases is not more than 3 in one organ, in the presence of a multi-organ lesion.
5. The total number of distant metastases is no more than 5.
6. Life expectancy of more than 6 months for brain metastases (GPA-score)
7. The possibility of SBRT for all distant metastases, in accordance with the criteria specified in the study design.
8. Making decisions on the inclusion of a patient in the study protocol based on the results of an interdisciplinary consultation consisting of an oncologist, a chemotherapist and a radiotherapist.
9. Signed informed consent

Exclusion Criteria:

1. 3-4 points on the WHO/ECOG scale of assessment of the general condition of the patient
2. The complete response of all foci to the chemotherapy.
3. Distant metastases only in the brain, without damage to bones and other organs.
4. Brain metastasis of more than 3 cm in one dimension, requiring surgical treatment.
5. Distant metastasis in the brain stem and spinal cord.
6. The size of at least one distant metastasis is more than 5 cm.
7. Previously performed radiation therapy on one of the metastatic foci.
8. Metastatic lesion of the pleura, membranes of the brain or peritoneum.
9. The impossibility of CTT for all distant metastases, in accordance with the criteria specified in the study design.
10. Invasion into great vessels (aorta, carotid arteries, pulmonary arteries, etc.), organs of the digestive tract (esophagus, stomach, intestines), skin.
11. Compression of the spinal cord by distant metastasis according to instrumental studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | At approximately end of year 1, 2,3 (study completion)
  Time period before cancer progression after the treatment, assessed in months
Time before the current drug line change | At approximately the end of years 1, 2, 3 (study completion)
  Time period before the indication for drug therapy alteration after the treatment, assessed in months

SECONDARY OUTCOMES:
Acute side effects | At approximately the end of months 1, 2, 3 (treatment completion)
  Local changes of tissues after the treatment, assessed in accordance to CTCAE v5.0
Late side effects | At approximately the end of years 1, 2, 3 (study completion)
  Local changes of tissues after the treatment, assessed in accordance to CTCAE v 5.0
Overall survival | At approximately the end of years 1, 2, 3 (study completion)
  Time period before patient death after the treatment, assessed in years
Local metastasis control | At approximately the end of years 1, 2, 3 (study completion)
  Time period before irradiated targets relapse, assessed in years/months
Quality of life Assessed with the Functional Assessment via EQ-5D (EuroQolGroup Scale) and The Numerical Rating Pain Scale | At approximately the end of month 1, 2, 3, 6, 12 (study completion)
  1. Functional Assessment via EQ-5D (EuroQolGroup Scale). The scale will be applied before treatment, and after the treatment at month 1, 2, 3, 6, 12 The system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems (a 1-digit number that expresses the level). The EQ visual-analogue records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can image' and 'The worst health you can image'. It will be used as a quantitative measure of health outcome that reflects the patient's own judgement.
  2. in case of painful targets The Numerical Rating Pain Scale will be applied before and after the treatment at month 1, 2, 3, 6, 12 . Score 0 (no pain) to 10 (maximal pain)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Gordon, Principal Investigator — A. Tsyb Medical Radiological Research Center
Locations (1):
- A. Tsyb Medical Radiological Research Center, Obninsk, Kaluga Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request from the principal investigator for researchers, who meet the criteria for access to confidential data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: unlimited
Access Criteria: informed consent for personal data non-disclosure